CLINICAL TRIAL: NCT06799039
Title: Pilot Trial of Xylitol for C. Difficile De-Colonization in Patients With Inflammatory Bowel Disease
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jessica Ravikoff Allegretti, Jessica R. Allegretti, MD, MPH, FACG, AGAF, Principle Investigator, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000210
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Inflammatory Bowel Disease (IBD); Clostridioides Difficile Infection
Keywords: C. Difficile; Decolonization; IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Clostridium Infections | interventions — Xylitol

STUDY DESIGN:
Intervention Model Description: Dose Finding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dose Finding Cohort (Experimental): One of five consecutively increasing dosing groups of xylitol
  Interventions: Drug: Xylitol
- Observational Cohort (No Intervention): Participants will be assessed for rates of spontaneous decolonization, stool sample testing and IBD scoring.

INTERVENTIONS:
Drug: Xylitol — Xylitol is a sugar alcohol and considered a GRAS substance by the FDA. Patients will be consecutively enrolled into one of five dosing including 1g, 2g, 5g, 7g and 9g.
  Arms: Dose Finding Cohort

SUMMARY:
This 3+3 dose escalation pilot trial will assess the safety and efficacy of xylitol as an oral therapeutic for decolonization of C. difficile in the Inflammatory Bowel Disease (IBD) patient population.

DETAILED DESCRIPTION:
Participants with confirmed IBD diagnosis who are scheduled for an outpatient colonoscopy for any reason at Brigham and Women's Hospital will be eligible for enrollment. Participants will be screened for C. difficile colonization via colonic wash sampling during colonoscopy. Participants may only have inactive or mild IBD at the time of the colonoscopy to be eligible.

Eligible participants will be initially enrolled in the observational cohort until there are 39 subjects enrolled. Participants in the observational cohort will be assessed at Week 1, 4 and 8, following confirmation of colonization. Participants will only be assessed for stool sample testing, IBD scoring and occurrence of CDI.

The subsequent participants who meet eligibility criteria will be enrolled into one of five consecutively increasing dosing groups of xylitol. The dose A treatment arm will receive a daily dose of 1 gram of xylitol for 7 days. The dose B treatment arm will receive a daily dose of 2 grams of xylitol for 7 days. The dose C treatment group will receive a daily dose of 5 grams of xylitol for 7 days. The dose D treatment group will receive a daily dose of 7 grams of xylitol for 7 days. The dose E treatment group will receive a daily dose of 9 grams of xylitol for 7 days. Participants will end dosing at day 7 but monitoring will continue through to week 8.

Participants in the will be assessed through week 8 for the primary outcome, determining the maximum tolerated dosage of xylitol. C. difficile decolonization will be assessed through week 8. Participants will also receive weekly phone call for assessment of symptoms and tolerability through week 8. In addition, secondary efficacy outcomes including IBD disease activity and development of CDI will be evaluated at week 8, and week 26. Participants will also be followed through week 26 for long-term safety, efficacy, and clinical outcomes. Disease activity and symptoms will be recorded from informed consent through the week 26 trial visit.

The primary outcome, determining the maximum tolerated dose of xylitol at week 8 will be confirmed via adverse event reporting. Additional C. difficile testing will be done at week 26.

The study will prospectively enroll between 15 and 30 adult participants at a single center. Participants that experience intolerable adverse events will be withdrawn from the study and will be considered treatment failures.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Male or female ≥ 18 years of age
3. IBD diagnosis (CD, UC or indeterminant Colitis will be permitted)
4. Inactive or mild IBD (HBI score ≤ 4; Partial Mayo score ≤ 4)
5. Presenting for outpatient colonoscopy or clinic appointment

Exclusion Criteria:

1. Unable to provide consent.
2. Patients with previous colectomy, ostomy, J-pouch, or previous colon surgery (excluding appendectomy)
3. Unable to complete study procedures.
4. Chronic use of antibiotics.
5. Inability or unwillingness to swallow capsules.
6. Allergy to xylitol.
7. Currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Efficacy of Xylitol | 8 weeks
  Incidence of Treatment Emergent Adverse Events (TEAEs) through Week 8
C. Diff Decolonization | 8 weeks
  Proportion of patients decolonized of C. difficile at Week 8

SECONDARY OUTCOMES:
Biomass of C. Difficile | 8 weeks
  Change in biomass of C. difficile in patients at Week 8
Effect of C. difficile decolonization on Inflammatory Bowel Disease (IBD) clinical outcomes | 26 weeks
  Change in IBD clinical score at Week 8 and Week 26. IBD clinical scores are used to assess IBD patient symptoms. The assessments are separated between scores for Ulcerative Colitis (UC) and Crohn's Disease (CD). The Harvey Bradshaw Index (HBI) is a clinical assessment for IBD patients with Crohn's disease while Partial Mayo Score is a clinical assessment for Ulcerative Colitis. The scores will be collected at study visit in form of a survey. The HBI score can vary but a score above 8 or 9 is considered severe disease activity. The Partial Mayo Score can range from 0 to 9 and a score above 7 is considered severe disease activity. A decrease in score from baseline to follow-up timepoints is indicative of improved IBD patient symptoms.
C. Difficile infection surveillance | 26 weeks
  Incidence of patients developing C. Difficile Infection through Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Allegretti, MD MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No